CLINICAL TRIAL: NCT05873101
Title: Comparison Of Effectiveness of Mobilization With Movement (MWM) and Kelternborn Treatment Technique to Increase ROM, Reducing Pain in Patient of ACL Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/539
Record Dates: First submitted 2023-03-18; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Movement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilization With Movement (MWM) (Other)
  Interventions: Diagnostic Test: Mobilization With Movement (MWM)
- Kelternborn Treatment Technique (Experimental)
  Interventions: Diagnostic Test: Kelternborn Treatment Technique

INTERVENTIONS:
Diagnostic Test: Mobilization With Movement (MWM) — Mobilization With Movement
  Arms: Mobilization With Movement (MWM)
Diagnostic Test: Kelternborn Treatment Technique — Kelternborn Treatment Technique
  Arms: Kelternborn Treatment Technique

SUMMARY:
To determine the Comparison Of Effectiveness of Mobilization With Movement (MWM) and Kelternborn Treatment Technique to Increase ROM, Reducing Pain in Patient of ACL Reconstruction

ELIGIBILITY:
Inclusion Criteria:

* • Subjects with age group between 20 to 60 years with sedentary lifestyle were included.

  * Both males and females were included.
  * Patients with diagnosed Tight hamstrings having knee extension less than 160º with the hip at 90º flexion.
  * Patients with decreased ROM at the knee joint.
  * Patients with reduced straight leg raise.
  * Patients with pain in posterior compartment of thigh.
  * Asymptomatic patients will be included.

Exclusion Criteria:

* • Patients with prolapsed disc were excluded.

  * Patients with lower extremity injuries (strain, sprain, ligament injuries, etc.) in last 6 months were excluded.
  * Patients with severe hamstring injury either acute or chronic were excluded.
  * Patients with visual acute swelling in the region of hamstring muscle
  * Patients with fracture of any type and area.
  * Patients with dislocations or subluxations present were excluded.
  * Patient recommended for TKR of knee joint.
  * Patients with any neurological disease like lumbar/cervical herniation, polyneuropathy, scoliosis etc.)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Goniometer (Range of Motion) | 6 Months
Visual Analog Scale ( VAS) | 6 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Superior University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No